CLINICAL TRIAL: NCT06538324
Title: Response to an Intervention With Omega-3 Fatty Acids on Lipid and Inflammatory Profiles in Overweight and Obese Individuals With Hypertriglyceridemia in Valdivia, Chile (RIO - Study)
Brief Title: Response to an Intervention With Omega-3 (RIO - Study)
Acronym: RIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad San Sebastián (Other)
Responsible Party: Principal Investigator, Viviana Sandoval, Researcher at the University San Sebastian, Universidad San Sebastián
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: CEC -USS N°42-24
Record Dates: First submitted 2024-07-10; First posted 2024-08-05 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-06

CONDITIONS: Overweight; Hypertriglyceridemia
Keywords: Omega-3 fatty acids; Lipid profile; Inflammatory profile; Postprandial TG response
MeSH Terms: conditions — Overweight; Hypertriglyceridemia | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, double - blind, crossover study.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The principal investigator will have exclusive access to the randomization code, which specifies the order of administration (either starting with HOSO or omega-3). This code is generated by an external statistician. The PI will ensure that the identical boxes containing capsules (both HOSO and Omega-3) are marked only with an Identification (ID). The randomization code will remain unknown to the participant, care provider, and outcomes assessor until after the primary outcome data has been analyzed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Marine Omega-3 fatty acid supplement (Experimental): Participants will be randomized to either star to receive a capsule/day with omega-3 fatty acid from 1g Nannochloropsis sp. microalga (250 mg of EPA) for 6 weeks. Followed by a wash-out period of 10 weeks.
  Interventions: Dietary Supplement: Omega-3
- High-oleic sunflower oil (HOSO) containing no EPA or other omega-3 fatty acid (Placebo Comparator): Participants will be randomized to either star to receive a placebo capsule/day with the same weight of high oleic sunflower oil -HOSO (with no EPA or other omega-3 fatty acid content), for 6 weeks. Followed by a wash-out period of 10 weeks.
  Interventions: Dietary Supplement: HOSO

INTERVENTIONS:
Dietary Supplement: Omega-3 — Dietary Supplement: Omega-3 In the marine Omega-3 fatty acid period, the participants will receive a capsule with 250 mg of EPA per day during 6 weeks.
  Arms: Marine Omega-3 fatty acid supplement
Dietary Supplement: HOSO — Dietary Supplement: HOSO In the HOSO period, the participants will receive a capsule with the similar weight of HOSO per day during 6 weeks.
  Arms: High-oleic sunflower oil (HOSO) containing no EPA or other omega-3 fatty acid

SUMMARY:
The RIO-Study project is a randomized, controlled, double-blind, crossover trial aimed at determining the effectiveness of omega-3 fatty acids at nutritional doses on lipid metabolism and inflammation in overweight and obese individuals with hypertriglyceridemia in Chile.

DETAILED DESCRIPTION:
The study will include 40 participants (each participant will serve as their own control) aged 18-65, with 25-34.9 kg/m2 BMI and fasting triglycerides (TG) of 100-215 mg/dL. The intervention consists of 250 mg EPA from algae oil versus high oleic sunflower oil (HOSO) for 6 weeks each, after a 10-week washout period, the treatments will be switched for another 6 weeks, considering four visits during the whole study. The main outcomes to be evaluated are serum triglyceride levels, expression of target genes in peripheral blood mononuclear cells (PBMCs), low-grade inflammation biomarkers, and very low-density lipoprotein (VLDL) atherogenic properties. The study also analyzes background diet, chrononutrition, and physical activity aspects. Results are expected to provide new insights into the effects of nutritional doses of omega-3 in the Chilean population, particularly on fasting and postprandial triglyceride metabolism and cardiovascular disease risk reduction.

Before and after each intervention period, fasting blood samples will be collected. On each visit day, participants will consume a standardized breakfast (three slices of white bread with butter and jam), and postprandial blood samples will be taken at 0, 2, 4, and 6 hours to measure triglycerides and other lipid parameters.

The study will assess:

1. Serum triglyceride levels in fasting and postprandial states
2. Expression of target genes Peroxisome proliferator-activated receptor alpha (PPARα) and Sterol regulatory element binding protein-1 (SREBP1c) in peripheral blood mononuclear cells (PBMCs) at fasting (0h) and postprandial (4h) states
3. Levels of low-grade inflammation biomarkers Tumor Necrosis Factor-Alpha (TNFα) and Interleukin 6 ( IL-6) at fasting (0h) and postprandial (4h) states
4. Very low-density lipoprotein (VLDL) atherogenic properties in the fasting state Additionally, the investigators will collect data on chrononutrition, physical activity, and energy drink intake to understand their impact on lipid metabolism. Anthropometric measurements and bioimpedance analysis will be performed at each visit.

The study will collaborate with international partners for specialized analyses, including gene expression studies and VLDL atherogenic properties assessment.

This comprehensive approach aims to provide new insights into the effects of nutritional doses of omega-3 fatty acids on lipid metabolism and inflammation in the Chilean population, with a particular focus on postprandial triglyceride metabolism and cardiovascular disease risk reduction.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18 and 65 years old, male and female.
* Body mass index (BMI) between 25 - 34,9 kg/m2.
* Fasting triglycerides between 100-215 mg/dL (1.13-2.43 mmol/L).

Exclusion Criteria:

* Unable to give informed consent.
* If you consume Omega-3 (you must stop consumption at least 10 weeks prior).
* Normal or Obesity Nutritional Status. Large weight variation (>10%) in the last 3 months.
* Triglycerides > 215 mg/dL.
* Blood pressure > 140/90 mmHg.
* Uncontrolled metabolic and chronic diseases (reference parameters for the disease in question will be considered).
* Pregnant women or those who are breastfeeding.
* Allergy or intolerance to gluten, milk protein and/or lactose, or any ingredient in the capsules (omega-3, oleic acid oil).
* Use of medications that affect lipid metabolism: Fibrates. (Statins will be allowed only if the treatment has been ongoing for over 3 months).
* Blood donation two months before or during the study period.
* Excessive alcohol consumption (>3 cans of beer per day)
* Taking anticoagulants.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-07-30 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Fasting TG (mg/dL) | up to 6 weeks
  Baseline serum levels of circulating triglycerides

SECONDARY OUTCOMES:
Postprandial TG (mg/dL) | up to 6 weeks
  Triglyceride concentration (mg/dL) measured by enzymatic colorimetric assay at baseline (fasting) and at 2, 4, and 6 hours after consumption of a standardized 50 g fat meal.
Change in mRNA expression levels of lipid metabolism genes in Peripheral Blood Mononuclear Cells (PBMCs) | up to 6 weeks
  Fold change in mRNA expression of genes of lipid metabolism in PBMCs at 0h and 4h, measured by RT-qPCR
Change in concentrations (pg/mL) of pro-inflammatory cytokines TNF-α and IL-6 | up to 6 weeks
  Serum concentrations (pg/mL) of tumor necrosis factor-alpha (TNF-α) and interleukin-6 (IL-6) measured by enzyme-linked immunosorbent assay (ELISA) at fasting (0h) and 4 hours postprandial following a standardized test meal
Fasting serum Low-Density Lipoproteins, High-Density Lipoproteins, Very Low-Density Lipoproteins (mg/dL) | up to 6 weeks
  Fasting levels before and after intake of omega-3 or HOSO
Fasting plasma glucose concentration (mg/dL) | up to 6 weeks
  Fasting levels before and after intake of omega-3 or HOSO

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad San Sebastián, Valdivia, Los Ríos Region, Chile

REFERENCES:
- See also: RIO-Study web site — https://www.rio-study.com/